CLINICAL TRIAL: NCT05045261
Title: ANRS HB07 IP-Cure-B Proof of Concept (PoC) Clinical Trial. Educating the Liver Immune Environment Through TLR8 Stimulation Followed by NUC Discontinuation
Acronym: IP-CURE-B
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: EUCLID Clinical Trial Platform (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS HB07 IP CURE B; 2020-004376-18 (EudraCT Number)
Record Dates: First submitted 2021-08-04; First posted 2021-09-16 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- A - Standard of care NUC (No Intervention): Patients will continue their standard of care NUC treatment
- B - NUC discontinuation (Experimental): Patients will stop their NUC treatment 28 weeks after enrolment
  Interventions: Drug: Discontinuation of NUC treatment in arms B and C
- C - NUC discontinuation after SLGN treatment (Experimental): Patients will take from enrolment
  * their standard of care NUC treatment for 28 weeks then stop
  * 3mg SLGN weekly for 24 weeks then stop
  Interventions: Drug: administration of SLGN in arm C; Drug: Discontinuation of NUC treatment in arms B and C

INTERVENTIONS:
Drug: administration of SLGN in arm C — administration of 3mg SLGN weekly for 24 weeks in arm C
  Arms: C - NUC discontinuation after SLGN treatment
Drug: Discontinuation of NUC treatment in arms B and C — NUC treatment will be stopped after 28 weeks in arms B and C
  Arms: B - NUC discontinuation; C - NUC discontinuation after SLGN treatment

SUMMARY:
The ANRS HB07 IP-cure-B study is a proof of concept Phase II clinical trial in HBeAg negative virally suppressed non-cirrhotic CHB patients. It will explore whether stopping NUC or stopping NUC after SLGN administration can increase the rate of HBsAg decline compared to standard of care CHB treatment.

DETAILED DESCRIPTION:
Epidemiology

Chronic hepatitis B (CHB) is a major public health care issue worldwide and one of the principal causes of chronic liver disease, cirrhosis and hepatocellular carcinoma (HCC). Liver cancer is the third leading cause of cancer deaths globally, with the highest burden of disease found in regions where HBV is endemic.

WHO estimates that in 2015, 257 million people were living with CHB infection (defined as hepatitis B surface antigen [HBsAg]-positivity) representing a worldwide prevalence of 3.9%, with considerable geographic variability. In 2015, hepatitis B resulted in an estimated 887,000 deaths, mostly from cirrhosis and HCC, placing it among the top 20 causes of mortality worldwide.

As of 2016, 27 million people (10.5% of all people estimated to be living with hepatitis B) were aware of their infection, while 4.5 million (16.7%) of the people diagnosed were on treatment.

Standard-of-care for CHB treatment

Nucleos(t)ide (NUC) analogs, administered orally, are the standard of care treatment for CHB, providing durable suppression of viral replication, defined by the decline of serum HBV DNA below the lower limit of quantification of diagnostic assays. NUC induced viral suppression, which is observed in the vast majority of patients (> 95%), results in long-term clinical benefits with a reduced risk of liver complications, i.e. decreased risk of: i) liver fibrosis progression, ii) hepatic decompensation in patients with pre-existing cirrhosis, and iii) HCC development. However, treatment with NUC rarely results in clearance of HBsAg and seroconversion to HBsAb even after long-term administration. In highly selected patient populations, the rate of HBsAg loss can reach 10% after 5 years of Tenofovir disoproxil fumarate (TDF) administration.

New treatment options that enhance rates of HBsAg clearance with or without seroconversion are needed. Such treatments will allow patients to discontinue life-long oral antiviral therapy and provide an option for a functional cure with a finite duration of treatment. A therapy with a finite duration of treatment is expected to be applicable to a broader population of chronically infected patients with HBV, including those that are not currently considered eligible for treatment with available therapies by the current clinical practice guidelines. For example, immunotolerant patients and inactive carriers do not fall within the current treatment indications. Different treatment strategies aimed to increase the HBsAg loss rates, either different regimens of currently available medications or regimens including new direct acting antivirals or immune modulators, are being explored.

The host immune response to HBV infection plays a pivotal role in whether acute infection is resolved or becomes chronic. It is also pivotal for control of intrahepatic viral cccDNA, which acts as a viral minichromosome. Individuals who are able to clear HBV infection spontaneously following an acute infection display a vigorous, polyclonal, HBV-specific CD8+ and CD4+ T cell response and maintain trace amounts of intrahepatic cccDNA. In contrast, CHB is associated with a limited and dysfunctional CD8+ T cell response, impaired natural killer (NK) cell antiviral function, the persistence of transcriptionally active cccDNA, and active viral replication. Novel approaches under investigation to achieve functional cure include direct inhibition of the viral replication cycle, targeting of cccDNA, and the stimulation of antiviral immune responses.

Rationale for the trial

The ANRS HB07 IP-cure-B study is a proof of concept Phase II clinical trial in HBeAg negative virally suppressed non-cirrhotic CHB patients. It will explore whether stopping NUC or stopping NUC after SLGN administration can increase the rate of HBsAg decline compared to standard of care CHB treatment. Exploratory analyses will help elucidate whether modifications in the liver immune environment are responsible for HBsAg decline.

The ANRS HB07 IP-Cure-B PoC clinical trial will be conducted in virally-suppressed HBeAg-negative CHB subjects to minimize safety risks and maximize efficacy benefits associated with SLGN. Because they achieve long-term viral suppression under NUC therapy, these subjects have lower levels of HBV DNA in the serum as well as lower expression of HBV antigens, especially HBsAg. A virally suppressed population may have a higher chance of responding to SLGN, as suggested by the observation that immune responsiveness of CHB patients is improved in patients who are on chronic suppressive antiviral therapy with low HBsAg levels. Of note, only subjects with excellent hepatic reserve, i.e. non-cirrhotic patients with normal liver function tests, will be included in this study to further maximize safety. Moreover, in virally suppressed patients with normal liver function, any alteration of liver enzymes will be easier to interpret.

A similar line of reasoning applies for the stopping NUC strategy, since patients with lower HBsAg levels have a higher chance of losing HBsAg after NUC cessation. The enrolment of patients without extensive liver fibrosis, per EASL clinical practice guidelines, will also minimize the risk of severe ALT flares after NUC withdrawal.

Hypothesis of the trial

The hypothesis tested in this trial is built on previous clinical investigations of the stopping NUC strategy and of SLGN administration in patients with CHB.

Thus, the investigators expect that the modification of the liver immune environment induced by SLGN administration should amplify the modifications of the immune responses induced by NUC withdrawal and lead to a restoration of effective intrahepatic innate immunity and HBV-specific T cell responses. In this PoC clinical trial, the investigators will explore, in HBeAg negative virally suppressed HBV patients, whether a TLR8 agonist (SLGN) treatment followed by NUC discontinuation can increase the rate of HBsAg decline.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HBeAg negative CHB on documented NUC for ≥ 3 years with HBV DNA LLOQ by local assay by polymerase chain reaction (PCR) documented at least annually over the last 3 years. NUC can include only tenofovir disoproxil fumarate (TDF), tenofovir alafemanide fumarate (TAF) or entecavir,
2. HBsAg ≥ 100 IU/mL but < or = 3,000 IU/mL at screening,
3. Male and female subjects aged 18 to 70 years (inclusive) at the day of screening,
4. Ultrasound, computed tomography (CT) scan, or magnetic resonance imaging (MRI) within 6 months of screening date with no evidence of hepatocellular carcinoma (HCC),
5. No evidence of advanced fibrosis or cirrhosis at screening: elastography (Fibroscan) value ≤ 9 kPa and ultrasonography without any sign of cirrhosis and platelets ≥ 150x109/L,
6. No evidence of advanced fibrosis or cirrhosis before the onset of NUC therapy,
7. HBV DNA < 20 IU/mL at screening,
8. ALT levels within the normal range of the local lab (< ULN) at screening,
9. Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of IMP. If the urine pregnancy test is positive, a follow-up serum test is required for confirmation,
10. Women of childbearing potential must agree to use a highly effective method of contraception from screening throughout the study period and for 7 days after the last dose of study drug. Men with female partners who are of childbearing potential must agree that they or their partners will use a highly effective method of contraception from screening throughout the study period and for 7 days after the last dose of study drug.

    1. Women of childbearing potential are sexually mature women who have not undergone bilateral oophorectomy or hysterectomy; or who have not been postmenopausal (ie, who have not menstruated at all) for at least 1 year.
    2. Highly effective methods of contraception not using hormonal contraceptives will be intrauterine device, tubal sterilization, Essure microinsert system; male partner sterilization; or total abstinence from heterosexual intercourse, when this is the preferred and usual lifestyle of the subject. Note: The double-barrier method (eg, synthetic condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), periodic abstinence (such as calendar, symptothermal, post-ovulation), withdrawal (coitus interruptus), lactational amenorrhea method, and spermicide only are not acceptable as highly effective methods of contraception.
11. Screening Electrocardiogram (ECG) without clinically significant abnormalities and with QTcF interval (QT corrected using Fridericia's formula) ≤ 450 msec for males and ≤ 470 msec for females,
12. Must be willing and able to comply with all study requirements,
13. Must have the ability to understand and sign a written informed consent form (ICF),
14. Participant covered by Health Insurance (when requested by local regulations)

Exclusion Criteria:

1. Any history of decompensation of liver disease including history of ascites, encephalopathy and gastrointestinal bleeding,
2. Any sign of oesophageal and/or gastric varices,
3. Laboratory parameters not within defined thresholds:

   1. White blood cells < 4,000 cells/μL (< 4.0×109/L);
   2. Hemoglobin < 11 g/dL (< 110 g/L) for females, < 13 g/dL (< 130 g/L) for males;
   3. Platelets < 130,000 per μL (< 130×109/L);
   4. Albumin < 3.5 g/dL (< 35 g/L);
   5. International normalized ratio (INR) > 1.5;
   6. Total bilirubin > 1.2 mg/dL (> 20.52 μmol/L). Note: subjects with an elevated indirect bilirubin and known Gilbert's disease can be included if direct bilirubin is within normal limits.
   7. Alpha-fetoprotein (AFP) > 20 ng/mL;
   8. Creatinine clearance (using the Cockcroft-Gault method) < 60 mL/min;
4. Co-infection with hepatitis C virus (HCV) (antibodies anti-HCV positive), human immunodeficiency virus type 1 (HIV-1) (antibodies anti-HIV positive) or hepatitis D virus (HDV) (antibodies anti-HDV positive),
5. Evidence or history or suspicion of hepatocellular carcinoma,
6. Malignancy within 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc). Note: subjects under evaluation for possible malignancy are not eligible.
7. Significant cardiovascular, pulmonary, or neurological disease,
8. Received solid organ or bone marrow transplant,
9. Received within 3 months of screening or expected to receive prolonged therapy with immunomodulators (eg, corticosteroids, anti-TNF) or biologics (eg, monoclonal antibody, IFN),
10. Subjects currently taking medication(s) that are transported through organic anion transporting polypeptide 1 (OATP1) including, but not limited to: atazanavir, rifampin, cyclosporine, eltrombopag, gemfibrozil, lopinavir/ritonavir, and saquinavir,
11. Concomitant treatment with the following medications (if taken within 21 days prior the baseline visit through the end of treatment plus 7 days)/diet:

    1. Hematologic stimulating agents (eg, erythropoiesis-stimulating agents; granulocyte colony stimulating factor [GCSF]; and thrombopoietin [TPO] mimetics),
    2. Potent CYP3A4 inhibitors or inducers, including but not limited to antifungals (fluconazole, ketoconazole…), antibiotics (telithromycin, rifabutin, rifampicin…), St. John's Wort, grapefruit juice, anticonvulsants (carbamazepine, phenobarbital, phenytoin…) etc,
    3. Immunosuppressant (except short term use of prednisone as a steroid burst [≤ 1 week of use]) and cytotoxic medications,
12. Known hypersensitivity or resistance to study drugs or formulation excipients,
13. Diagnosis of autoimmune disease (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune hepatitis, sarcoidosis, psoriasis of greater than mild severity, autoimmune uveitis), poorly controlled diabetes mellitus, significant psychiatric illness, severe chronic obstructive pulmonary disease, hemoglobinopathy, retinal disease, or immunosuppressed patients,
14. Use of another investigational agent within 6 months of screening and during the whole duration of the trial,
15. Current alcohol or substance abuse judged by the Investigator to potentially interfere with compliance,
16. Females who are breastfeeding, pregnant or may wish to become pregnant during the study,
17. Female subjects unwilling to refrain from egg donation and in vitro fertilization during and until at least 7 days after the last study drug dose. Male subjects unwilling to refrain from sperm donation during and until at least 7 days after the last study drug,
18. Any medical condition that, in the opinion of the investigator, could interfere with evaluation of the study objectives or safety of the subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy : Percentage of subjects with ≥ 1.0 log10 IU/mL decline of HBsAg at week 76 | Week 76
  percentage of subjects with ≥ 1.0 log10 IU/mL decline of HBsAg at week 76 compared to baseline

SECONDARY OUTCOMES:
Efficacy : Percentage of subjects with HBsAg ≥ 0.3 log10 IU/mL decline | Weeks 12, 24, 28, 36, 48, 76
  Percentage of subjects with HBsAg ≥ 0.3 log10 IU/mL decline at weeks 12, 24, 28, 36, 48, 76 compared to baseline
Efficacy : Percentage of subjects with HBsAg ≥ 0.5 log10 IU/mL decline | Weeks 12, 24, 28, 36, 48, 76
  Percentage of subjects with HBsAg ≥ 0.5 log10 IU/mL decline at weeks 12, 24, 28, 36, 48, 76 compared to baseline76 compared to baseline
Efficacy : Percentage of subjects with HBsAg ≥ 1.0 log10 IU/mL decline | Weeks 12, 24, 28, 36, 48, 76
  Percentage of subjects with HBsAg ≥ 1.0 log10 IU/mL decline at weeks 12, 24, 28, 36, 48 compared to baseline
Efficacy : Percentage of subjects with HBsAg < 100 IU/mL | Weeks 12, 24, 28, 36, 48, 76
  Percentage of subjects with HBsAg < 100 IU/mL at weeks 12, 24, 28, 36, 48, 76Percentage of subjects with HBsAg < 100 IU/mL at weeks 12, 24, 28, 36, 48, 76
Efficacy : Percentage of subjects with HBsAg < 10 IU/mL | Weeks 12, 24, 28, 36, 48, 76
  Percentage of subjects with HBsAg < 10 IU/mL at weeks 12, 24, 28, 36, 48, 76
Efficacy : Percentage of subjects with HBsAg loss | Weeks 12, 24, 28, 36, 48, 76
  Percentage of subjects with HBsAg loss at weeks 12, 24, 28, 36, 48, 76 and time to HBsAg loss since baseline
Efficacy : Percentage of subjects with HBsAb seroconversion | Weeks 12, 24, 28, 36, 48, 76
  Percentage of subjects with HBsAb seroconversion at weeks 12, 24, 28, 36, 48, 76 and time to HBsAb seroconversion
Efficacy : Changes in serum HBsAg, HBcrAg, HBV RNA and HBV DNA levels in log10 IU/mL | Weeks 12, 24, 28, 36, 48, 76
  Changes in serum HBsAg, HBcrAg, HBV RNA and HBV DNA levels in log10 IU/mL from baseline to weeks 12, 24, 28, 36, 48, 76
safety/tolerance : Percentage of subjects reporting a grade 3 or 4 AE | Up to week 76
  Percentage of subjects reporting a grade 3 or 4 AE
safety/tolerance : Percentage of all grade AEs | Up to week 76
  Percentage of all grade AEs
safety/tolerance : Percentage of subjects with ALT flares | Up to week 76
  Percentage of subjects with ALT flares at each time point (ALT flares defined as ≥ 10 x ULN)
safety/tolerance : Percentage of subjects with NUC treatment re-initiated | Up to week 76
  Percentage of subjects in whom NUC treatment has been re-initiated.
quality of life of the participants | at baseline, weeks 28 and 76
  To assess and compare health-related quality of life, measured using the EuroQol-5Dimension-5Levels(EQ-5D-5L) utility score

CONTACTS AND LOCATIONS:
Overall Officials: Fabien ZOULIM, MD, Principal Investigator — Hepatology Department, Hospices Civils de Lyon
Locations (8):
- France (4):
  - Hepatology Department, Hospices Civils de Lyon, Lyon
  - Hepato-gastroenterology department, Hôpital Saint-Joseph, Marseille
  - Service d'Hépato-gastroentérologie, Hôpital de Brabois, Nancy
  - Service d'Hépato-gastroentérologie Hôpital Pitié Salpêtrière, Paris
- Department of Internal Medicine Clinic for Internal Medicine II - Gastroenterology, Hepatology, Endocrinology and Infectiology, Universitat Klinikum in Freiburg, Freiburg im Breisgau, Germany
- Italy (2):
  - Gastroenterology and Hepatology Division, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Department of General and Specialized Medical AreaAzienda Ospedaliera, University Hospital of Parma, Parma
- Internal Medicine and Hepatology, Vall d'Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Research projects may be submitted and evaluated by the Trial Scientific committee for scientific relevance. If the projects receives a favorable opinion, a data sharing agreement shall be signed.
  Participants will be informed of any further research project and will have the opportunity to refuse the use of their data